CLINICAL TRIAL: NCT02625831
Title: Association Between the Presence of Autoantibodies Targeting Ficolin-3 and Active Nephritis in Patients With Systemic Lupus Erythematosus
Brief Title: Anti-ficolin-3 Autoantibodies in Lupus Nephritis
Acronym: ficolupus
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 1841851v0
Record Dates: First submitted 2015-11-13; First posted 2015-12-09 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: ficolin-3; anti-ficolin-3 antibodies; lupus nephritis; Lupus Erythematosus, Systemic; biomarker
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Biological Oxygen Demand Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — one serum sample per patient.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SLE patients: 165 SLE patients. Subgroup : 77 with active lupus and 88 in disease remission. in the active subgroup : 36 with lupus nephritis and 41 without.
  Biological analysis were performed.
  Interventions: Other: Biological analysis
- healthy patients: 48 healthy patients. Biological analysis were performed.
  Interventions: Other: Biological analysis

INTERVENTIONS:
Other: Biological analysis — Biological analysis :
  * ficolin-3
  * anti-ficolin 3 antibodies
  * anti-C1q antibodies
  Other Names: Biological analysis on pre-existing serum collection

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease characterized by the production of multiple autoantibodies. Antibodies against Ficolin-3 were previously identified in the sera of some SLE patients, but their prevalence and significance have not been yet investigated. The aims of this study were to determine the prevalence of anti-ficolin-3 antibodies among SLE patients and to investigate their potential as diagnostic and/or prognostic biomarkers in SLE.

In this retrospective study, clinical data were obtained from medical files and blood samples were selected from preexisting biological collection. SLE patients (n=165) were informed and did not objected, they were matched to healthy controls (n=48). Disease activity was determined according to the SLEDAI score. Anti-ficolin-3, anti-dsDNA and anti-C1q antibodies levels were measured in sera by ELISA. First, a highly significant difference was found in the anti-ficolin-3 levels between SLE patients and healthy subjects. Anti-ficolin-3 antibodies were detected as positive in 58 of 165 (35%) SLE patients. The titer of anti-ficolin-3 antibodies was correlated with the SLEDAI score (p<0.0001). The presence of anti-ficolin-3 antibodies was associated with anti-C1q and anti-dsDNA antibodies. Regarding associations with clinical manifestations, only the presence of active lupus nephritis was significantly associated with the presence of anti-ficolin-3 antibodies (p=0.0001). This association with renal involvement was higher with anti-ficolin-3 antibodies than with other auto-antibodies. Interestingly, the combination of anti-ficolin-3 and anti-C1q antibodies demonstrated higher specificity than any other traditional biomarker.

These results suggest that anti-ficolin-3 could be useful for the diagnosis of active nephritis in SLE patients.

DETAILED DESCRIPTION:
For this retrospective study, a brief summary should be enough.

ELIGIBILITY:
165 SLE patients

Inclusion Criteria:

* Age: ≥ 18 years old
* Patients with lupus diagnostic criteria (ACR1997)

Exclusion Criteria:

* Pregnant women
* Patient with known evolutive cancer

  48 healthy patients matched in age and sex with one or several SLE patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: SLE patients were studied from medical data files of the Departments of Internal Medicine (Grenoble University Hospital, France) and Nephrology (Conception University Hospital, Marseille, France). For SLE patients, clinical and biological manifestations as well as treatments received and disease activity evaluated using the SLE Disease Activity Index (SLEDAI) at the time of sampling were recorded. SLE patients were divided into subgroups as described in group section.
Sampling Method: Non-Probability Sample
Enrollment: 213 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Anti-ficolin-3 antibodies presence in SLE patients | measured at day of inclusion = T0.
  Anti-ficolin-3 antibodies in SLE patients, considered positive if superior than 70 arbitrary units.
  This study have a single visit approach with serum collection so every outcome is measured at T0, which is the only visit for the patient.

SECONDARY OUTCOMES:
Correlation of anti-ficolin-3 antibodies with anti-DNA antibodies in SLE patients | measured at day of inclusion = T0.
  This study have a single visit approach with serum collection so every outcome is measured at T0, which is the only visit for the patient.
Correlation of anti-ficolin-3 antibodies with anti-C1q antibodies in SLE patients | measured at day of inclusion = T0.
  This study have a single visit approach with serum collection so every outcome is measured at T0, which is the only visit for the patient.
Correlation of anti-ficolin-3 antibodies with lupus activity (SLEDAI score) in SLE patients | measured at day of inclusion = T0.
  This study have a single visit approach with serum collection so every outcome is measured at T0, which is the only visit for the patient.
Anti-ficolin-3 antibodies presence in SLE patients with active nephritis | measured at day of inclusion = T0.
  This study have a single visit approach with serum collection so every outcome is measured at T0, which is the only visit for the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Chantal DUMESTRE-PERARD, PhD, Principal Investigator — University Hospital Grenoble, FRANCE

IPD SHARING:
Plan to Share IPD: Undecided
sub-study still in progress. Further analysis is needed before sponsor can decide his Policy of sharing individual data for this research.

REFERENCES:
- [Background] Andersen T, Munthe-Fog L, Garred P, Jacobsen S. Serum levels of ficolin-3 (Hakata antigen) in patients with systemic lupus erythematosus. J Rheumatol. 2009 Apr;36(4):757-9. doi: 10.3899/jrheum.080361. Epub 2009 Feb 4. PMID 19208603
- [Background] Herrmann M, Voll RE, Zoller OM, Hagenhofer M, Ponner BB, Kalden JR. Impaired phagocytosis of apoptotic cell material by monocyte-derived macrophages from patients with systemic lupus erythematosus. Arthritis Rheum. 1998 Jul;41(7):1241-50. doi: 10.1002/1529-0131(199807)41:73.0.CO;2-H. PMID 9663482
- [Background] Honore C, Hummelshoj T, Hansen BE, Madsen HO, Eggleton P, Garred P. The innate immune component ficolin 3 (Hakata antigen) mediates the clearance of late apoptotic cells. Arthritis Rheum. 2007 May;56(5):1598-607. doi: 10.1002/art.22564. PMID 17469142
- [Background] Liphaus BL, Kiss MH. The role of apoptosis proteins and complement components in the etiopathogenesis of systemic lupus erythematosus. Clinics (Sao Paulo). 2010 Mar;65(3):327-33. doi: 10.1590/S1807-59322010000300014. PMID 20360925
- [Background] Orbai AM, Truedsson L, Sturfelt G, Nived O, Fang H, Alarcon GS, Gordon C, Merrill J, Fortin PR, Bruce IN, Isenberg DA, Wallace DJ, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke AE, Aranow CB, Manzi S, Urowitz MB, Gladman DD, Kalunian KC, Costner MI, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, Van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS, Petri M. Anti-C1q antibodies in systemic lupus erythematosus. Lupus. 2015 Jan;24(1):42-9. doi: 10.1177/0961203314547791. Epub 2014 Aug 14. PMID 25124676
- [Background] Yoshizawa S, Nagasawa K, Yae Y, Niho Y, Okochi K. A thermolabile beta 2-macroglycoprotein (TMG) and the antibody against TMG in patients with systemic lupus erythematosus. Clin Chim Acta. 1997 Aug 29;264(2):219-25. doi: 10.1016/s0009-8981(97)00078-8. No abstract available. PMID 9293379
- [Background] Sato N, Ohsawa I, Nagamachi S, Ishii M, Kusaba G, Inoshita H, Toki A, Horikoshi S, Ohi H, Matsushita M, Tomino Y. Significance of glomerular activation of the alternative pathway and lectin pathway in lupus nephritis. Lupus. 2011 Nov;20(13):1378-86. doi: 10.1177/0961203311415561. Epub 2011 Sep 5. PMID 21893562
- [Background] Kuraya M, Ming Z, Liu X, Matsushita M, Fujita T. Specific binding of L-ficolin and H-ficolin to apoptotic cells leads to complement activation. Immunobiology. 2005;209(9):689-97. doi: 10.1016/j.imbio.2004.11.001. PMID 15804047
- [Background] Lacroix M, Dumestre-Perard C, Schoehn G, Houen G, Cesbron JY, Arlaud GJ, Thielens NM. Residue Lys57 in the collagen-like region of human L-ficolin and its counterpart Lys47 in H-ficolin play a key role in the interaction with the mannan-binding lectin-associated serine proteases and the collectin receptor calreticulin. J Immunol. 2009 Jan 1;182(1):456-65. doi: 10.4049/jimmunol.182.1.456. PMID 19109177
- [Background] Takahashi R, Tsutsumi A, Ohtani K, Goto D, Matsumoto I, Ito S, Wakamiya N, Sumida T. Anti-mannose binding lectin antibodies in sera of Japanese patients with systemic lupus erythematosus. Clin Exp Immunol. 2004 Jun;136(3):585-90. doi: 10.1111/j.1365-2249.2004.02477.x. PMID 15147364